CLINICAL TRIAL: NCT07270133
Title: Longitudinal Natural History Study of Retinal Function in Eyes of Patients With Diabetes
Acronym: AR
Status: Not yet recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Protocol AR; UG1EY014231 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinal Disease
MeSH Terms: interventions — Visual Acuity; Visual Fields; Contrast Sensitivity; Electroretinography; Light; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Non-diabetic controls: Aged-matched people without a diagnosis of diabetes. At least one eye must be eligible without retinal pathology.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Reading Speed; Diagnostic Test: Visual Field testing; Diagnostic Test: Contrast sensitivity; Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states; Diagnostic Test: Ultrawide field-color photograph; Diagnostic Test: Ultrawide field-Fluorescein angiogram; Diagnostic Test: Optical coherence tomography; Other: Optical coherence tomography- Angiography
- Subclinical (No diabetic retinopathy on the diabetic retinopathy severity scale): Eyes of patients with a diagnosis of diabetes, Diabetic Retinopathy Severity Scale = 10, and no diabetic macular edema. Lower limit on duration of disease for Type 1 is 5 years, for Type 2 is 1 year
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Reading Speed; Diagnostic Test: Visual Field testing; Diagnostic Test: Contrast sensitivity; Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states; Diagnostic Test: Ultrawide field-color photograph; Diagnostic Test: Ultrawide field-Fluorescein angiogram; Diagnostic Test: Optical coherence tomography; Other: Optical coherence tomography- Angiography
- Minimal to Mild non-proliferative diabetic retinopathy: Eyes of patients with a diagnosis of diabetes, Diabetic Retinopathy Severity Scale = 20-35, and no center-involved diabetic macular edema
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Reading Speed; Diagnostic Test: Visual Field testing; Diagnostic Test: Contrast sensitivity; Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states; Diagnostic Test: Ultrawide field-color photograph; Diagnostic Test: Ultrawide field-Fluorescein angiogram; Diagnostic Test: Optical coherence tomography; Other: Optical coherence tomography- Angiography
- Moderate non-proliferative diabetic retinopathy: Eyes of patients with a diagnosis of diabetes, Diabetic Retinopathy Severity Scale = 43-47, and no center-involved diabetic macular edema
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Reading Speed; Diagnostic Test: Visual Field testing; Diagnostic Test: Contrast sensitivity; Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states; Diagnostic Test: Ultrawide field-color photograph; Diagnostic Test: Ultrawide field-Fluorescein angiogram; Diagnostic Test: Optical coherence tomography; Other: Optical coherence tomography- Angiography
- Severe non-proliferative diabetic retinopathy: Eyes of patients with a diagnosis of diabetes, Diabetic Retinopathy Severity Scale = 53, and no center-involved diabetic macular edema
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Reading Speed; Diagnostic Test: Visual Field testing; Diagnostic Test: Contrast sensitivity; Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states; Diagnostic Test: Ultrawide field-color photograph; Diagnostic Test: Ultrawide field-Fluorescein angiogram; Diagnostic Test: Optical coherence tomography; Other: Optical coherence tomography- Angiography
- Proliferative diabetic retinopathy: Eyes of patients with a diagnosis of diabetes, Diabetic Retinopathy Severity Scale > 60, and no center-involved diabetic macular edema
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Reading Speed; Diagnostic Test: Visual Field testing; Diagnostic Test: Contrast sensitivity; Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states; Diagnostic Test: Ultrawide field-color photograph; Diagnostic Test: Ultrawide field-Fluorescein angiogram; Diagnostic Test: Optical coherence tomography; Other: Optical coherence tomography- Angiography

INTERVENTIONS:
Diagnostic Test: Visual Acuity — Visual Acuity measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent of <20/800). Higher scores indicate better visual acuity, and lower scores indicate worse visual acuity
  Other Names: Early treatment diabetic retinopathy study visual acuity ETDRS
Diagnostic Test: Reading Speed — The MNREAD (Minnesota Low-Vision Reading) test is a standardized test that measures reading performance in people with normal or impaired vision.
  Other Names: MNREAD (Minnesota Low-Vision Reading)
Diagnostic Test: Visual Field testing — The objectiveFIELD Analyzer is a perimetry tool that measures visual fields using electroencephalography-based brain responses to flickering light. Higher sensitivity = better function, Lower sensitivity (more negative deviations from normal) = worse function; Global indices (MD, PSD-like values) indicate overall field loss and pattern of damage.
  Other Names: objectiveFIELD analyzer
Diagnostic Test: Contrast sensitivity — A clinical device that utilizes the quick Contrast Sensitivity Function (qCSF) methodology to assess visual function. The qCSF method is a Bayesian adaptive algorithm designed to efficiently estimate a patient's contrast sensitivity across a wide range of spatial frequencies. Higher curve / higher AULCSF = better contrast sensitivity (normal vision). Lower curve / lower Area Under the Log Contrast Sensitivity Function = reduced contrast sensitivity (seen in early AMD, glaucoma, diabetic retinopathy, etc.).
  Other Names: AST Manifold qCSF
Diagnostic Test: Electroretinography (ERG) and pupillography in light- and dark-adapted states — The RETeval® is a portable, handheld electroretinography (ERG) and visual evoked potential (VEP) device. It enables clinicians to assess the retinal and optic nerve.
  Other Names: RETeval device
Diagnostic Test: Ultrawide field-color photograph — Ultrawide field color photography is a high-resolution, wide-angle retinal imaging technique that captures both central and peripheral retina in natural color. Grading is typically based on the Diabetic Retinopathy Severity Scale or DRSS, which is a standardized grading scale from 10 (no DR) to 85 (severe PDR)
  Other Names: UWF-Photo
Diagnostic Test: Ultrawide field-Fluorescein angiogram — a high-resolution, wide-angle retinal vascular imaging technique that allows clinicians to see both central and peripheral retina blood flow, detect ischemia, leakage, and neovascularization, and guide diagnosis and treatment
  Other Names: UWF-FA
Diagnostic Test: Optical coherence tomography — non-invasive retinal imaging tool that produces detailed cross-sectional images. Disease-specific grading systems (like macular thickness for DME or RNFL thickness for glaucoma) are used to quantify severity and monitor progression
  Other Names: OCT
Other: Optical coherence tomography- Angiography — non-invasive, dye-free imaging method that maps retinal and choroidal vasculature, allowing both qualitative and quantitative assessment of microvascular health. Quantitative metrics like vessel density, perfusion, FAZ size, and non-perfusion area serve as functional "scales" for disease severity and progression.
  Other Names: OCT-A

SUMMARY:
A considerable hurdle to the development of novel, more effective therapies for diabetic retinal disease is the limited number of primary endpoints available for use in regulatory trials. Current endpoints necessitate long trial durations and a greater number of participants to show efficacy. Thus, a better understanding of the structural and functional changes in the retina occurring in people with diabetes is essential for developing primary endpoints and validating surrogate and clinical endpoints.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with Type 1 or Type 2 diabetes or non-diabetic control patients
* Best corrected visual acuity 20/32 or better (Snellen) (≥74 ETDRS letters)
* Meets criteria for one of the defined observational groups below
* Able and willing to provide informed consent

Key Exclusion Criteria:

* Ocular or systemic condition, aside from diabetes mellitus (DM), that is likely to affect the assessment of DRSS, DME, or the functioning of the neural retina
* Previous treatment of any kind for diabetic retinopathy or DME
* Any condition that may preclude adequate imaging of the macula (e.g. dense cataract or other media opacity, ptosis)
* History of rhegmatogenous retinal detachment or macular hole
* History of vitrectomy
* Intraocular surgery (including cataract surgery) within 4 months prior to enrollment or anticipated within the next 6 months
* Requiring treatment for DR/DME in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals must meet all of the inclusion criteria and none of the exclusion criteria to be eligible to participate in the study. The potential study participant must have at least one eye meeting the inclusion criteria, but participants may have both eyes eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Does the performance of the objectiveFIELD Analyzer at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  The objectiveFIELD Analyzer is a perimetry tool that measures visual fields using electroencephalography-based brain responses to flickering light. Higher sensitivity = better function, Lower sensitivity (more negative deviations from normal) = worse function; Global indices (MD, PSD-like values) indicate overall field loss and pattern of damage.
Does the performance of the Contrast sensitivity (AST Manifold qCSF) at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  A clinical device that utilizes the quick Contrast Sensitivity Function (qCSF) methodology to assess visual function. The qCSF method is a Bayesian adaptive algorithm designed to efficiently estimate a patient's contrast sensitivity across a wide range of spatial frequencies. Higher curve / higher AULCSF = better contrast sensitivity (normal vision). Lower curve / lower Area Under the Log Contrast Sensitivity Function = reduced contrast sensitivity (seen in early AMD, glaucoma, diabetic retinopathy, etc.).
Does the performance of the Electroretinography (ERG) at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  The RETeval® is a portable, handheld electroretinography (ERG) and visual evoked potential (VEP) device. It enables clinicians to assess the retinal and optic nerve.
Does the performance of the Ultrawide field-color photograph at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  Ultrawide field color photography is a high-resolution, wide-angle retinal imaging technique that captures both central and peripheral retina in natural color. Grading is typically based on the Diabetic Retinopathy Severity Scale or DRSS, which is a standardized grading scale from 10 (no DR) to 85 (severe PDR)
Does the performance of the Ultrawide field-Fluorescein angiogram at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  A high-resolution, wide-angle retinal vascular imaging technique that allows clinicians to see both central and peripheral retina blood flow, detect ischemia, leakage, and neovascularization, and guide diagnosis and treatment
Does the performance of the Optical coherence tomography at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  A non-invasive retinal imaging tool that produces detailed cross-sectional images. Disease-specific grading systems (like macular thickness for DME or RNFL thickness for glaucoma) are used to quantify severity and monitor progression
Does the performance of the Optical Coherence Tomography- Angiography at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  A non-invasive, dye-free imaging method that maps retinal and choroidal vasculature, allowing both qualitative and quantitative assessment of microvascular health. Quantitative metrics like vessel density, perfusion, FAZ size, and non-perfusion area serve as functional "scales" for disease severity and progression.
Does the performance of Visual Acuity at baseline worsen as the Diabetic Retinopathy Severity Score increases | 4 Years
  Visual Acuity measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent of <20/800). Higher scores indicate better visual acuity, and lower scores indicate worse visual acuity